CLINICAL TRIAL: NCT04834115
Title: Efficacy of Ivermectin in Outpatients With Non-severe COVID-19: A Randomized Controlled Trial
Brief Title: Efficacy of Ivermectin in Outpatients With Non-severe COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Nacional de Asunción (Other)
Collaborators: Consejo Nacional de Ciencias y Tecnologia, Paraguay (Unknown); Ministerio de Salud Pública y Bienestar Social, Paraguay (Unknown); Centro de información y recursos para el desarrollo, Paraguay (Unknown); Centro para el Desarrollo de la Investigación Científica, CEDIC, Paraguay (Unknown); Instituto Desarrollo, Paraguay (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PINV20-387
Record Dates: First submitted 2021-03-28; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Covid19; Coronavirus Infection
Keywords: Ivermectin; Communicable Diseases; Respiratory Tract Infections
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Communicable Diseases; Respiratory Tract Infections | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: This is a double blind, randomized controlled trial with two parallel groups that evaluates the efficacy of ivermectin in reducing hospitalization in outpatients with COVID-19.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin (Experimental): Ivermectin 200mcg/kg single dose, maximum dose 18mg
  Interventions: Drug: Ivermectin Tablets
- Placebo (Placebo Comparator): Inactive medication tablets indistinguishable from ivermectin tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ivermectin Tablets — Oral ivermectin at a one time dose
  Arms: Ivermectin
Other: Placebo — Oral placebo at a one time dose
  Arms: Placebo

SUMMARY:
This is a randomized controlled trial to evaluate the efficacy of ivermectin in reducing the risk of progression to severe disease and hospitalizations in COVID-19 patients.

DETAILED DESCRIPTION:
This is a randomized controlled trial to evaluate the efficacy of ivermectin in COVID-19 outpatients reducing the risk of progression to severe disease.

Patients with COVID-19 infection are randomized to receive a single dose of 200mcg/kg of ivermectin or a placebo.

The randomization code is generated by the trial statistician. The allocation is made after fulfilment of both inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnostic RT-qPCR or antigen test for SARS-CoV-2
* Symptomatic patients with up to 8 days from the onset of symptoms, and asymptomatic cases with up to 5 days of positive test for SARS-CoV-2.
* Patients who agree to participate in the study by signing the informed consent.

Exclusion Criteria:

* Patients with severity criteria defined in the Coronavirus Disease Epidemiological and Laboratory Surveillance Guide (Version 3/11/2020)
* Pregnant or breastfeeding women
* Women of childbearing age and without commitment to use contraceptive methods during the study time.
* Inability to complete the study
* Current treatment with drugs known to interact with ivermectin
* Known intolerance to ivermectin, its derivate or any of its excipients.
* Patients with known Child-Pugh C liver disease
* Patients with prior ivermectin consumption in the 10 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with hospitalization criteria | 30 days
  Proportion of patients with hospitalization criteria at day 30

SECONDARY OUTCOMES:
Proportion of patients with COVID-19 signs and symptoms | 14 days
  Proportion of patients with COVID-19 signs and symptoms up to day 14
Proportion of cohabitants who had COVID-19 after the index case | 30 days
  Proportion of cohabitants who had COVID-19 after the index case up to day 30
Drug-related adverse events | 30 days
  Proportion of patients with ivermectin adverse events up to day 30
Levels of IgG for SARS-CoV-2 | 30-60 days
  Quantitative levels of IgG for SARS-CoV-2 measured by ELISA immunoassay

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Ciencias Médicas - Universidad Nacional de Asunción, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No
The investigators will publish the results to compare data with other studies with ivermectin and SARS-CoV-2 infection.

REFERENCES:
- [Background] Lopez-Medina E, Lopez P, Hurtado IC, Davalos DM, Ramirez O, Martinez E, Diazgranados JA, Onate JM, Chavarriaga H, Herrera S, Parra B, Libreros G, Jaramillo R, Avendano AC, Toro DF, Torres M, Lesmes MC, Rios CA, Caicedo I. Effect of Ivermectin on Time to Resolution of Symptoms Among Adults With Mild COVID-19: A Randomized Clinical Trial. JAMA. 2021 Apr 13;325(14):1426-1435. doi: 10.1001/jama.2021.3071. PMID 33662102
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Background] Chaccour C, Ruiz-Castillo P, Richardson MA, Moncunill G, Casellas A, Carmona-Torre F, Giraldez M, Mota JS, Yuste JR, Azanza JR, Fernandez M, Reina G, Dobano C, Brew J, Sadaba B, Hammann F, Rabinovich R. The SARS-CoV-2 Ivermectin Navarra-ISGlobal Trial (SAINT) to Evaluate the Potential of Ivermectin to Reduce COVID-19 Transmission in low risk, non-severe COVID-19 patients in the first 48 hours after symptoms onset: A structured summary of a study protocol for a randomized control pilot trial. Trials. 2020 Jun 8;21(1):498. doi: 10.1186/s13063-020-04421-z. PMID 32513289
- See also: National Council of Science and Technology, Paraguay — https://datos.conacyt.gov.py/proyectos/pdf/3449